CLINICAL TRIAL: NCT05892809
Title: Effect of an Incubator Cover on Term and Preterm Neonates' Vital Signs: a Prospective Randomized Study
Brief Title: Effect of an Incubator Cover on Term and Preterm Neonates' Vital Signs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Behice Ekici, Assistant Professor, PhD, Maltepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MaltepeUniversity
Record Dates: First submitted 2023-04-30; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Neonatal Disease; Nursing Caries
Keywords: term; preterm; vital signs; incubator cover
MeSH Terms: conditions — Infant, Newborn, Diseases; Premature Birth

STUDY DESIGN:
Intervention Model Description: A Pretest-Posttest Repeated Measures Design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- With incubator cover group and without incubator cover (Other): The incubator cover was covered while the neonate was lying in the incubator. Vital signs were measured at 0th, 15th, and 30th minutes.
  Interventions: Other: use an incubator cover

INTERVENTIONS:
Other: use an incubator cover — Vital signs of term and preterm newborns were measured separately and with and without an incubator cover.

SUMMARY:
The aim of this study is to evaluate the effect of an incubator cover on the vital signs of term and preterm neonates hospitalized in a neonatal intensive care unit. Methods: 91 neonates presenting to a neonatal intensive care unit who met the inclusion criteria were included in the study. Vital signs of neonates were measured with and without incubator cover. Measurements were performed three times (0th, 15th, and 30th minute).

DETAILED DESCRIPTION:
Term and preterm are exposed to many stimuli during their stay in the neonatal intensive care unite (NICU). These stimuli; operation and alarm sounds of devices, continuous and high level ambient lighting. These stimuli can cause deviations in the physiological indicators of newborns, and hearing and vision loss. The aim of this study is to evaluate the effect of an incubator cover on the vital signs of term and preterm neonates hospitalized in a neonatal intensive care unit. Methods: This study is a prospective repeated measure pretest-posttest repeated-measures design. 91 term and preterm newborns who were hospitalized in the neonatal intensive care unit and met the inclusion criteria were included in this study.

Neonates were admitted to the study if they satisfied all of the following criteria: (1) term and preterms, (2) admitted to NICU, (3) clinically stable, (4) verbal and written consent from the parent. Term and preterm neonates were randomized into two groups (term group = 44, and preterm group = 47 neonates). Vital signs of both groups were measured with and without incubator cover. Measurements were performed three times (0th, 15th, and 30th minute).

ELIGIBILITY:
Inclusion Criteria:

* Parents giving verbal and written consent,
* Hospitalized in the II. Level NICU
* Those born at 38-42 weeks of gestation
* Those born at 24-38 weeks of gestation
* Newborns with a body weight of 1500-2500 grams

Exclusion Criteria:

* Having life-threatening health problems

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Measurement and monitoring of newborn's pulse rate | The change in the newborn's heart rate within 30 minutes was monitored and measured.
  Physiological parameters of newborns will be evaluated. Multi-parameter monitor will be used for pulse rate, The newborn's heart rate per minute was measured.
  Vital signs of term and preterm will be measured without and with incubator cover. Vital signs of newborns will be measured three times. These measurements will be made at 0th, 15th, and 30th minutes. The medians of the measurement results will be taken and interpreted according to the reference range of the physiological measurement parameters.
Measurement and monitoring of newborn's respiratory rate | The change in the newborn's respiratory rate within 30 minutes was monitored and measured.
  Physiological parameters of newborns will be evaluated. Multi-parameter monitor will be used for respiratory rate, The respiratory rate of the newborn per minute was measured.
  Vital signs of term and preterm will be measured without and with incubator cover. Vital signs of newborns will be measured three times. These measurements will be made at 0th, 15th, and 30th minutes. The medians of the measurement results will be taken and interpreted according to the reference range of the physiological measurement parameters.
Measurement and monitoring of newborn's oxygen saturation | The change in the newborn's oxygen saturation within 30 minutes was monitored and measured.
  Physiological parameters of newborns will be evaluated. Multi-parameter monitor will be used for oxygen saturation, The oxygen saturation of the newborn was measured.
  Oxygen saturation will be evaluated in %. Vital signs of term and preterm will be measured without and with incubator cover. Vital signs of newborns will be measured three times. These measurements will be made at 0th, 15th, and 30th minutes.The medians of the measurement results will be taken and interpreted according to the reference range of the physiological measurement parameters.
Measurement and monitoring of newborn's body temperature | The change in the newborn's body temperature within 30 minutes was monitored and measured.
  Physiological parameters of newborns will be evaluated. Multi-parameter monitor will be used for oxygen saturation, The body temperature of the newborn was measured.
  Body temperature will be evaluated in degrees Celsius. Vital signs of term and preterm will be measured without and with incubator cover. Vital signs of newborns will be measured three times. These measurements will be made at 0th, 15th, and 30th minutes.
  The medians of the measurement results will be taken and interpreted according to the reference range of the physiological measurement parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Kenan Çetin, Nurse, Principal Investigator — Neonatal Intensive Care Unit
Locations (1):
- Siverek State Hospital, Sanliurfa, Siverek, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No